CLINICAL TRIAL: NCT04028401
Title: Optimization of Skin Preparation to Reduce Cutibacterium Acnes Colonization in Superficial and Deep Samples During Prosthetic Shoulder Surgery in Male Patients
Acronym: OPRICA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC19_0042
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cutibacterium Acnes Infection
MeSH Terms: interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 % benzoyl peroxide topical treatment (Experimental): Application of 5% benzoyl peroxide
  Interventions: Drug: 5% benzoyl peroxide
- No topical treatment (No Intervention): No intervention

INTERVENTIONS:
Drug: 5% benzoyl peroxide — Application of 5% benzoyl peroxide during 5 days before the procedure
  Arms: 5 % benzoyl peroxide topical treatment

SUMMARY:
Infections on joint replacements remain one of the most serious complications of orthopaedic surgery. Despite improvements in skin preparation and antibiotic prophylaxis procedures, the risk of infection of joint prosthesis is still high, particularly for shoulder prostheses, especially in men. One of the bacteria most often involved in post-operative infections for shoulder prosthesis is Cutibacterium acnes (CA). This bacterium is one of the predominant bacteria in pilosebaceous units. Eradication of this micro-organism remains difficult despite the techniques used in the preoperative phase.

The objective of this protocol is to evaluate the efficacy of applying a 5% benzoyl peroxide topical during the 5 days preceding the procedure in the surgical skin incision area, which is based on local acne treatment, on the reduction of the CA bacterial load in the dermis of the approach to shoulder arthroplasty in men.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, Adult patients,
* Patient without a history of surgical intervention on the operated shoulder,
* Patient managed for glenohumeral, partial (cup or anatomical hemi- arthroplasty) or total (anatomical or inverted) glenohumeral arthroplasty placement for primary osteoarthritis, or secondary to necrosis, massive rotator cuff tear or old fracture.
* Patients affiliated to a social security system
* Patients who have given their informed and written consent

Exclusion Criteria:

* Patient with arthroplasty for resumption of previous shoulder surgery or failure of arthroplasty
* Patient with arthroplasty for acute trauma
* Patient on immunosuppressantsimmunosuppressive drugs
* Patient with inflammatory rheumatism
* Patient with progressive cancer pathology
* Allergies or intolerances concerning the modalities of selected skin preparations (Povidone Iodine, hypersensitivity to benzoyl peroxide)
* Dermatological pathologies in the area to be treated
* Acne treatment in the area to be treated within four weeks before inclusion
* Patient without possible help from a third party for the application of Cutacnyl® 5% in the intervention group if necessary
* Major under guardianship
* Patient under the protection of justice
* Patient not covered by social security

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients in each group with a positive Cutibacterium acnes sample at the dermis. | Day 0

SECONDARY OUTCOMES:
Average number of positive intraoperative Cutibacterium acnes samples | Day 0
  samples taken at he cutaneous level before and after cutaneous antisepsis of the operating area before incision, fat and capsular.
Average number of positive Cutibacterium acnes skin samples before and after alcoholic surgical site antisepsis (5% alcoholic iodine povidone) in each of the two study groups | Day 0
Incidence of Cutibacterium acnes shoulder prosthesis infections up to 2 years after shoulder prosthesis implantation in both study groups | 2 years
Phylotype | Day 0
  Determination of phylotype by molecular typing by Multi-Locus Sequence Typing and Single-Locus Sequence Typing techniques and comparison of Cutibacterium acnes strains by molecular biology and characterization of antibiotic resistance
Cutibacterium acnes strains | Day 0
  Comparison of Cutibacterium acnes strains by molecular biology
Antibiotic resistance | Day 0
Evaluation of the skin tolerance of the topical application from the skin tolerance scale (irritation, erythema and desquamation), at the time of inclusion and at D0 | Day 0
  skin tolerance scale evaluates local tolerance (absent: 0, light:1, moderate: 2 severe:3), erythema (absent:0, light:1, moderate:2, severe:3, very severe:4) and desquamation (absent: 0, light: 1, moderate: 2, severe: 3, very severe: 4)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane CORVEC, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No